CLINICAL TRIAL: NCT05660928
Title: Control of Hypertension and diAbetes in MINas Gerais: Assessment of the Impact of Implementing a Multidimensional Strategy for Management of Patients With Systemic Arterial Hypertension and Diabetes Mellitus in Primary Care
Brief Title: Control of Hypertension and diAbetes in MINas Gerais
Acronym: CHArMING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Federal University of the Valleys of Jequitinhonha and Mucuri (Other); Medical Research Council (Other Government); University of Southampton (Other)
Responsible Party: Principal Investigator, Antonio Luiz Pinho Ribeiro, Professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 55598822.0.0000.5149
Record Dates: First submitted 2022-11-16; First posted 2022-12-21 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Arterial Hypertension; Diabetes Mellitus
Keywords: Hypertension; Diabetes mellitus; Telemedicine; Primary health care
MeSH Terms: conditions — Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Eighteen primary care centers will be randomized to the intervention arm, which consists of a multidimensional strategy, with a multidisciplinary approach, for the management of patients with hypertension and diabetes in the primary care setting. It is going to include:
  1. Telehealth tools: clinical decision support system for primary care professionals to support the care of patients with hypertension and diabetes; clinical decision support system to support community health agents (ACS), for use in home visits; asynchronous teleconsultations; telediagnosis for digital electrocardiogram and retinography reports; text messages to patients, to provide information, education, improve adherence to treatment and encourage patients to promote health;
  2. Continued education for health professionals;
  3. Strengthening the educational groups and promotion of lifestyle changes, with a focus on promoting healthy eating and reducing sedentary behavior.
  Interventions: Other: Multidimensional intervention
- Usual care (No Intervention): Seventeen primary care centers will be randomized to usual care.

INTERVENTIONS:
Other: Multidimensional intervention — Multidimensional intervention, with mutidisciplinary approach.
  Arms: Intervention

SUMMARY:
Hypertension and diabetes mellitus (DM) are highly prevalent in low and middle-income countries, and the proportion of patients with uncontrolled diseases is higher than in high income countries. Innovative strategies are required to surpass barriers of low sources, distance, and quality of healthcare. Our aim is to assess the uptake and effectiveness of the implementation of an integrated multidimensional strategy in the primary care setting, for the management of patients with hypertension and diabetes mellitus (DM) in Brazil. This is a scale up implementation study that has mixed-methods, and comprehends four steps: (1) needs assessment, including a standardized structured questionnaire and focus groups with healthcare practitioners; (2) baseline period, three months before the implementation of the intervention; (3) cluster randomized controlled trial (RCT) with a 12-month follow-up period; and (4) a qualitative study after the end of follow-up. The cluster RCT will randomize 35 centres to intervention (n= 18) or usual care (n= 17). Patients ≥18 years-old, with diagnosis of hypertension and/or DM, of five Brazilian cities in a resource-constrained area will be enrolled. The intervention consists of a multifaceted strategy, with a multidisciplinary approach, including telehealth tools (decision support systems, short message service, telediagnosis), continued education with an approach to issues related to the care of people with hypertension and diabetes in primary care, including pharmacological and non-pharmacological treatment and behavioural change. The project has actions focused on professionals and patients.

DETAILED DESCRIPTION:
This scale up implementation study has mixed-methods, and comprehends four steps: (1) needs assessment, (2) baseline period, (3) cluster RCT and (4) qualitative study. The RE-AIM planning and evaluation framework will be used in this research project, which includes: reach (R), efficacy (E), adoption (A), implementation (I), and maintenance (M). The Adaptation Framework might be used as well, in case adaptations need to be conducted during the intervention, taking into account the COVID-19 pandemic and possible new waves.

1. A standardized structured questionnaire will be developed with open questions about the physical and technological structure, human resources and challenges managing patients with hypertension and DM, in order to carry out a brief situational diagnosis.
2. A baseline period of three months will be established to assess the basal condition of patients. Individuals will be assessed for blood pressure and glycohemoglobin measurements; functional performance (2-minute step test); anthropometric measurements (weight, height, and waist circumference); physical inactivity; alcohol consumption; smoking; and food consumption markers.
3. A two-arm parallel cluster RCT will be conducted, with a baseline period of three months and a subsequent follow-up period of 12 months from the start of the intervention. To avoid possible contamination within the same primary care unit, randomization will take place at a primary care centre level: each centre will be randomized to the control or the intervention arm, rather than individual patients. Randomization will be performed by computer software and stratified by geographic location and municipality, to ensure balance between arms.
4. At the end of the cluster-randomized controlled trial, another qualitative study will be carried out using the FG technique, in order to assess barriers and suggestions for improvement of each component of the implemented multidimensional strategy.

To calculate the sample size, the investigators took into account the proportion of patients with controlled hypertension (33%) and DM (37%) observed at baseline in the pilot study (data not published), and an absolute increase of 6% in these proportions one year after the implementation of the intervention, with a power of 0.80, level of significance of 0.05 and intra cluster correlation coefficient of 0.026. The calculated sample was 34 primary care centres, 17 in each arm, with a minimum of 148 participants in each centre. As the total number of primary care centres in the five municipalities is 35, the investigators planned to include one extra unit in the intervention arm. Taking into account a drop out rate of up to 17.8%, the total number of included individuals will be 180.

ELIGIBILITY:
Inclusion Criteria:

Primary Health Care - Basic health unit with internet availability and complete team, including a Brazilian doctor or with a proficiency test in the Portuguese language.

Patients

- Adult patients (from 18 years-old), diagnosed with hypertension and/or DM, registered in the medical record.

Subproject cluster randomised controlled trial. All of the above criteria and the following additional criteria:

* Patients aged ≥ 18 years-old, with a diagnosis of hypertension and diabetes mellitus, registered in the medical record;
* Absence of contraindications to physical activity, according to the assistant physician's assessment;
* In intervention levels II and III, it will be a prerequisite that the participant has a smartphone.

Exclusion Criteria:

* Patients with terminal illness, with a life expectancy lower than 12 months according to the physician's evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5862 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Composite outcome of proportion of patients with controlled disease | 12 months
  (i) for hypertension, the proportion (%) of patients with systolic blood pressure (SBP) <140 mmHg and diastolic blood pressure (DBP) < 90 mmHg; (ii) for diabetes, the proportion (%) of patients with glycohemoglobin ≤ 7% if the age < 60 years, or < 8% if the age is ≥ 60 years; (iii) for those with both hypertension and diabetes, proportion (%) of patients with both diseases controlled.

SECONDARY OUTCOMES:
Proportion of patients with controlled hypertension | 12 months
  The proportion (%) of patients with systolic blood pressure (SBP) <140 mmHg and diastolic blood pressure (DBP) < 90 mmHg
Proportion of patients with controlled diabetes | 12 months
  The proportion (%) of patients with glycohemoglobin ≤ 7% if the age < 60 years, or < 8% if the age is ≥ 60 years
Change in blood pressure | 12 months
  The mean difference in delta SBP and DBP (mmHg) in patients with hypertension, when comparing the intervention and the control groups, in 12 months
Change in glycohemoglobin | 12 months
  The mean difference in delta glycohemoglobin (%) in patients with diabetes, when comparing the intervention and the control groups, in 12 months
Number of blood pressure measurements | 12 months
  Number of blood pressure measurements per patient with hypertension in 12 months
Number of glycohemoglobin measurements | 12 months
  Number of glycohemoglobin measurements per patient with diabetes in 12 months

OTHER OUTCOMES:
Percentage of patients who participated in group activities in 12 months. | 12 months
  Percentage of patients with hypertension and diabetes who participated at least once in group activities in 12 months.
Total follow-up time of patients | 12 months
  Time in months between the first consultation after enrollment and last consultation during the study period
Number of consultations during the follow-up time | 12 months
  Number of consultations with medical doctors and nurses during the follow-up time
Performance in the 2-minute standing gait test | 6 and 12 months
  The difference in the number of steps (delta from the beginning) in the 2-minute standing gait test within 6 months and 12 months.
Performance in the hand grip strength test | 6 and 12 months
  The difference in the hand grip strength measured by in kgf (delta from the beginning) within 6 months and 12 months.
Change in the body weight | 12 months
  The change in the body weight (kg) in the follow-up time
Change in the body mass index | 12 months
  The change in the body mass index in the follow-up time
Change in the waist circumference | 12 months
  The change in the waist circumference (cm) in the follow-up time
Program adherence | 12 months
  Total follow-up time (time between the first consultation after enrollment and last consultation); median time between medical and nurse consultations; number of consultations during follow-up time, number of groups conducted at each primary care centre during the follow-up; participation of patients at the educational groups; adherence to CDSS recommendations (intervention group only).

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Minas Gerais, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Derived] Fonseca SF, Ribeiro ALP, Cimini CCR, Soares TBC, Delfino-Pereira P, Nogueira LT, Moura RMF, Motta-Santos D, Ribeiro LB, Camargos MCS, Paixao MC, Pires MC, Batchelor J, Marcolino MS. Scale up of implementation of a multidimensional intervention to enhance hypertension and diabetes care at the primary care setting: A protocol for a cluster-randomized study in Brazil. Am Heart J. 2023 Aug;262:119-130. doi: 10.1016/j.ahj.2023.04.006. Epub 2023 Apr 11. PMID 37044364